CLINICAL TRIAL: NCT00750126
Title: Feasibility Study on Allogeneic Hematopoietic Stem Cell Transplantation Following Fludarabine-Busulfan-ALS-based Reduced-intensity Conditioning in Children With Hematological Malignancy or Solid Tumor Not Responding to Standard Therapy or for Which the Indication for Allograft is Maintained But Cannot be Carried Out Due to the Toxicity Involved in Myeloablative Conditioning.
Brief Title: Allogeneic Hematopoietic Stem Cell Transplantation
Acronym: RICE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Dr Catherine PAILLARD, CHU Clermont-Ferrand
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0039
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Solid Tumors; Hematologic Neoplasms
Keywords: Allograft; Children; malignancy; Reduced Intensity Conditioning; Fludarabin; Busulfex; Thymoglobulin
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasms | interventions — fludarabine; Busulfan; thymoglobulin

INTERVENTIONS:
Drug: Fludarabine, Busulfan, Thymoglobulin — study :
  * acute and/or chronic graft-versus-host reaction (incidence and severity) and immune reconstitution, post transplantation
  * the effectiveness of the protocol on tumor response
  * overall survival

SUMMARY:
To assess the engraftment of hematopoietic stem cells following reduced-intensity conditioning in children presenting with solid tumors or hematological malignancy by evaluating post-transplantation chimerism and hematological reconstitution.

To study acute and/or chronic graft-versus-host reaction (incidence and severity) and immune reconstitution, post-transplantation To study the effectiveness of the protocol on tumor response.

To study overall survival.

DETAILED DESCRIPTION:
Primary criterion

* Hematological reconstitution and chimerism post-transplantation

Secondary criteria

* Adverse effects, graft-related mortality at D90 and at 12 months, incidence and severity of acute and/or chronic GVH reactions
* Analysis of variations in post-transplantation immunological function profiles
* Median duration of response in therapy-responsive patients and median duration of stability in stabilized patients

ELIGIBILITY:
Inclusion Criteria:

* Patients aged less than 20 years old
* Lansky score > 60%
* Life expectancy greater than 2 months
* Diagnoses:

  3- Solid tumor or hematological malignancy remaining unresponsive to the reference strategies according to French best practices in pediatrics.

  4- Malignancies for which allografting is the recognized indication but is contraindicated with myeloablative conditioning.
* Usual criteria for allogeneic grafting (pre-graft profile)
* Having a HLA-identical sibling donor for HLA-A, HLA-B and HLA-DR antigens or a HLA mismatch on only one antigen, or having a 10/10 pheno-identical donor, or compatible cord blood.
* Signed informed consent

Exclusion Criteria:

* Patient presenting rapidly-progressive malignancy
* In cases where the potential donor is related, sibling presenting contraindication against hematopoietic stem cell donation
* Unable to sufficiently understand the treatment and its consequences, even after explanation

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-04; Primary Completion 2009-04 (Estimated); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Primary criterion - Hematological reconstitution and chimerism post-transplantation | post-transplantation

SECONDARY OUTCOMES:
Secondary criteria - Adverse effects, graft-related mortality at D90 and at 12 months, incidence and severity of acute and/or chronic GVH reactions | post-transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Paillard Catherine, Dr, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Paillard Catherine, Clermont-Ferrand, France